CLINICAL TRIAL: NCT06784076
Title: Establishing the Salience of Type 1 Interferon Pathway Blockade in the Central Mechanisms of SLE Related Fatigue
Acronym: EPIC
Status: Not yet recruiting | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Other Study IDs: GN23RH258
Record Dates: First submitted 2025-01-13; First posted 2025-01-20 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — anifrolumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood sample.
  Urine sample is also taken as part of pregnancy test for female participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Anifrolumab — Anifrolumab 300mg intravenous infusions administered as described in the EU SmPC
  Other Names: N/A (Not applicable)

SUMMARY:
Systemic Lupus Erythematosus (SLE) is a multi-system autoimmune disorder, characterised by activation of the interferon system. Of the multiple domains of this disease, patients identify fatigue as the most pervasive and disabling aspect. As many as 90% report significant levels of fatigue, a prevalence far in excess of that observed in the general population and most other chronic disorders. Moreover, its impact permeates all aspects of living as reflected by fatigue's strong relationship with impaired quality of life3 and work disability. Despite these substantial consequences, relatively little is known about this symptom and so the current dearth of accepted therapies is unsurprising. A better understanding of the underlying mechanisms of fatigue will be vital if efficacious interventions are to be developed in the future.

The investigators will recruit 25 SLE patients to achieve 20 full data sets. They will attend for a baseline 7T brain scan to primarily measure basal ganglia glutamate and then receive 5 months of a pharmacological blocker that antagonises type 1 interferon receptors before completing the study with a final 7T brain scan to undertake repeat measure of basal ganglia glutamate.

DETAILED DESCRIPTION:
Our epidemiological investigations of fatigue in autoimmune disease have identified strong associations with central nervous system factors such as mental health and cognitive dysfunctions, and the investigators have subsequently pioneered the application of advanced MRI brain methods in order to derive neurobiological mechanistic insights into fatigue. As a result, the investigators have implicated basal ganglia volume to be a key marker of fatigue severity. The basal ganglia has been considered pivotal in neuroimaging studies of fatigue across the chronic disease spectrum11 and fatigue is a defining clinical characteristic of basal ganglia disorders such as Parkinson's disease. Intriguingly, a 3 Tesla (3T) MRI spectroscopy study of Hepatitis C patients evidenced possible increases in basal ganglia glutamate concentrations following treatment with interferon α which in turn correlated with worsening reported levels of fatigue. Glutamate is the brain's foremost excitatory neurotransmitter. Pre-clinical experiments suggest that inflammatory cytokines can enhance extracellular glutamate levels through various mechanisms including decreasing activity of glutamate metabolising enzymes and reversing cellular efflux. The consequences of heightened glutamate include altered neuronal integrity and microglial activation. Correspondingly, it is notable that peripheral administration of interferon α in a mouse model induced both molecular and phenotypic activation in microglia.

Basal ganglia glutamate could be an important mediator of fatigue in diseases, such as SLE, which are underpinned by type 1 interferon pathway activation. However, until recently, it has not been possible to robustly investigate this possibility further in humans. Standard 3T MRI scanners fail to provide sufficient spectral resolution to distinguish glutamate from glutamine (a distinct metabolite) and so previous studies offer only preliminary evidence. The University of Glasgow now benefits from one of the few UK ultra-high field 7T MRI scanners to be embedded in a clinical research facility. The use of 7T rather than 3T MRS (Magnetic Resonance Spectroscopy) permits a highly resolved quantifiable glutamate signal within small subcortical regions due to higher Larmor frequency and improved chemical shift dispersion. The investigators have successfully applied single voxel MRS sequences at 7T to quantify glutamate in autoimmune disease, which enables the required precision to robustly measure glutatmate.

A downstream impact of any glutamate imbalance may be dysfunctional brain activity. Functional MRI (fMRI) leverages the differential magnetic strength of oxygenated and deoxygenated haemoglobin to generate a Blood Oxygen Level Dependent (BOLD) signal, a surrogate measure of brain activity. In autoimmune disease, the investigators have also related fatigue to enhanced fMRI connectivity to a number of brain regions, in particular the Dorsal Attention Network. Fatigue was also significantly associated with increased Default Mode Network to insula functional connectivity. This is the most reproducible biomarker of fibromyalgia, a chronic pain disorders that is defined by co-existing fatigue and is conspicuously prevalent in SLE where it is indeed a major predictor of fatigue.

These innovations in MRI imaging now allow us to opportunely use anifrolumab to pharmacologically block type 1 interferon receptors in order to test our hypothesis that blockade of the type 1 interferon pathway will lead to reductions in brain basal ganglia glutamate. This in turn will facilitate understanding of the mechanism of fatigue being caused in people with SLE.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years < 65 years
* Fulfilment of the 2019 ACR (American College of Rheumatology)/EULAR (European Alliance of Associations for Rheumatology) classification criteria for SLE
* Persistent (>3 months) and clinically significant fatigue (≥6 on numerical rating 0-10 scale measuring average level of fatigue during the past 7 days)
* Attainment of Lupus low disease activity state (LLDAS)

Exclusion Criteria:

* Inability to provide informed written consent
* Moderate or severe active SLE
* Severe active CNS (Central Nervous System) Lupus and Lupus Nephritis
* Contra-indications to anifrolumab
* History of malignancy
* History of recurrent infections or known risk factors for infection
* Active or chronic infection
* Concomitant biological therapies
* Hypersensitivity to anifrolumab or excipients
* Current treatment with a biologic medicine or monoclonal antibody (including B cell depleting therapies in the previous 52 weeks)
* Previous exposure to anifrolumab
* Contra-indications to MRI
* Pregnant or breast-feeding
* Females of child-bearing potential who do not agree to use an effective method of birth control until 12 weeks after the final study visit (See appendix 1).)
* Severe physical impairment (e.g. blindness, paraplegia)
* Medical or psychiatric conditions that in the judgement of the study personnel would preclude participation in the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: SLE Patients attending NHS Greater Glasgow & Clyde, NHS Lanarkshire, NHS Forth Valley, NHS Tayside and NHS Grampian rheumatology department with low disease activity state aged over 18 years less than75 years. The total number of participants will be 20.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-03-17 (Estimated); Primary Completion 2025-03-17 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Changes in basal ganglia glutamate levels | 0-18 weeks
  Changes in basal ganglia glutamate levels measured by 7T MRI following pharmacological blockade of type 1 interferon receptors in SLE .

SECONDARY OUTCOMES:
Changes in dorsal attention network (DAN) | 0-18 weeks
  Changes in dorsal attention network (DAN) as measured by 7T MRI
Changes in default mode network (DMN) - insula brain connectivity | 0-18 weeks
  Changes in default mode network (DMN) - insula brain connectivity as measured by 7T MRI

OTHER OUTCOMES:
Changes of fatigue as measured via Functional Assessment of Chronic Illness Therapy - Fatigue Scale | 0-18 weeks
  To describe any changes of fatigue in association with altered glutamate and brain functional connectivity using the Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-F).
  The FACIT-F scale consists of 13 items that assess the level of fatigue experienced by the respondent over the past 7 days. These items cover various aspects of fatigue, such as physical, emotional, and functional well-being.
  Each item is rated on a 5-point Likert scale, with response options ranging from "Not at all" (0) to "Very much" (4). The respondent selects the option that best describes their experience.
  The scores for each item are summed to create a total score. Some items are reverse-scored to ensure that higher scores consistently indicate better functioning and less fatigue. The total score can range from 0 to 52, with higher scores indicating less fatigue and better quality of life.
Changes of fatigue as measured via the Patient-Reported Outcomes Measurement Information System Fatigue Scale. | 0-18 weeks
  To describe any changes of fatigue in association with altered glutamate and brain functional connectivity using the Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Scale.
  The PROMIS Fatigue Scale includes a large item bank with questions related to fatigue. These questions cover various aspects of fatigue, such as its intensity, frequency, and impact on daily activities.
  Each question has five response options, usually ranging from "Not at all" to "Very much." These responses are scored on a scale from 1 to 5, with higher scores indicating greater fatigue.
Longitudinal modulation of the Type 1 Interferon Transcriptomic Signature in the Peripheral Immune Compartment | 0-18 weeks
  This outcome investigates the changes in the pattern of gene expression related to type 1 interferons over time in the immune cells found in the blood and other peripheral tissues. These changes will be measured as part of research blood samples in each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Basu, MD, PhD, Principal Investigator — neil.basu@glasgow.ac.uk